CLINICAL TRIAL: NCT04292795
Title: Effect of Shortwave Diathermy Versus Therapeutic Ultrasound on Medial Tibial Stress Syndrome Among Military Cadets
Brief Title: Effect of Shortwave Diathermy and Therapeutic Ultrasound on Medial Tibial Stress Syndrome Among Military Cadets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shifa Clinical Research Center (Other)
Responsible Party: Principal Investigator, Dr. Tahir Ramzan, Lecturer, Shifa Clinical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Applied_for_IRB
Record Dates: First submitted 2020-02-26; First posted 2020-03-03 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Medial Tibial Stress Syndrome
Keywords: Medial Tibial Stress Syndrome; Pain; Pain Syndrome; Cadets
MeSH Terms: conditions — Medial Tibial Stress Syndrome; Pain; Somatoform Disorders | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Intervention: Shortwave Diathermy Frequency: 27.12 MHz Time Duration: 10min Duration of Treatment: 4 weeks. Sessions per Week: 2 sessions per week
  Interventions: Device: Short wave diathermy
- Group B (Experimental): Intervention: Therapeutic Ultrasound Frequency: 1-3MHz Intensity: 0.2-1W/cm2 Time Duration: 10mins Duration of Treatment: 4 weeks Sessions per Week: 2 sessions per week
  Interventions: Device: Therapeutic Ultrasound

INTERVENTIONS:
Device: Therapeutic Ultrasound — The Intervention will be provided according to the set protocols used in previous literature.
  Arms: Group B
Device: Short wave diathermy — The Intervention will be provided according to the set protocols used in previous literature.
  Arms: Group A

SUMMARY:
Medial tibial stress syndrome (MTSS) also known as shin splints or tibial periostitis is a common injury in athletes and soldiers/cadets with incidences ranging between 4% and 35% in these populations . It is characterized by pain in the middle and lower end of tibia; the pain is usually elicited by practicing sports or other physical activities. The criteria for diagnosis for MTSS were established by Yates and White. Although the prognosis of MTSS is usually benign, it can evolve to chronicity and be disabling.

Several studies have demonstrated the effects of different medical treatment in athletes and cadets with MTSS. Study will correspond to the demonstration of treatment options for medial tibial stress syndrome that lie in the domain of Physical Therapy.

Therapeutic Ultrasound and Shortwave Diathermy.

DETAILED DESCRIPTION:
Primary objective of the study includes:

1. To determine the effect of Shortwave Diathermy on Medial Tibial Stress Syndrome among military cadets.
2. To determine the effect of Therapeutic Ultrasound on Medial Tibial Stress Syndrome among military cadets.
3. To compare the effects of Shortwave Diathermy and Therapeutic Ultrasound on Medial Tibial Stress Syndrome among military cadets.

study hypothesis is "Shortwave diathermy and Therapeutic Ultrasound are equally effective in Medial Tibial Stress Syndrome among military cadets.".

Study Design : Randomized Control trial Study Settings is Pakistan Military Academy Abbottabad. Sample Size: The sample size calculation is done through epitool to obtain a sample size ratio 1:1 for both treatment groups with Power of 0.8, Confidence interval of 0.95 and Variance = 5.

Mean of experimental group was 2.17 and mean of control group was 4.26 taken from the parent article.

Results obtained from epitool:

Total sample size: 36 Sample size per group: 18(each group) Sampling Technique: Non-probability Purposive Sampling- subjects will be recurited into the groups through sealed enveloped method.

Work Plan/Timeline for Participants:

Timeline for the participants will be one month after the approval of IRB form.

Follow ups:

There will be 2 follow ups per week for a period of 4 weeks.

Statistical Analysis:

Data will be analyzed on Statistical Package for Social Sciences (SPSS) version 21.

Descriptive Results:

* Quantitative data will be interpreted in terms of means and standard deviation whereas qualitative data will be presented in the form of frequencies and percentages.
* Quantitative data will be represented in form of histogram whereas qualitative data is shown in the form of bar charts and graphs.

Interferential Results:

* Data will be assessed for its normality by applying Shapiro-Wilk test and its value of 0.05 or lesser than that shows that the data is normally distributed at baseline and at the end of treatment.
* Parametric test will be used for normally distributed data whereas non parametric test would be applied for skewed sample or away from normality data.
* For comparison between two groups, Independent T Test (parametric) or Mann-Whitney Test(non-parametric) will be used both a baseline and at the end of sessions.
* For within the group comparison at intervals (baseline and post treatment), Pared T test (parametric) or Wilcoxon Rank Test (non-parametric) will be applied.

ADVERSE/SERIOUS ADVERSE EFFECTS / POTENTIAL HAZARDS:

No adverse effects are present in this study. Onsite clinical arrangements will be made available for subjective and objective assessment and for the treatment protocol as well. For this purpose portable modalities will be used which will be easy to transfer and operate. The total expenses required will be provided by the students themselves

No potential risk present to the participants or community as a whole

POTENTIAL BENEFIT TO THE PARTICIPANTS OR COMMUNITY AS WHOLE

1. Awareness will be provided regarding MTSS among community.
2. Long term complications leading to physical limitations and disability will be prevented.
3. Awareness regarding Physical Therapy treatment for MTSS will be provided

ELIGIBILITY:
Inclusion Criteria:

1. Age: 19-24 years
2. Gender: Male
3. Cadets diagnosed with Medial tibial stress syndrome according to Yates and White Criteria(3).

Exclusion Criteria:

1. Individuals having stress fractures or history of stress fractures.
2. Local infection or osteomyelitis.
3. Tumor in assessment region.
4. Compartment syndrome.
5. Musculoskeletal problems or other comorbidities.

Ages: 19 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Pre Numeric Pain Rating Scale (NPRS) | the outcome will be assessed at baseline (day zero).
  The outcome measure suitable for evaluating the severity of pain in medial tibial stress syndrome
Post-Numeric Pain Rating Scale (NPRS) | the outcome will be assessed at end of 4th week
  The outcome measure suitable for evaluating the severity of pain in medial tibial stress syndrome
Pre-Medial Tibial Stress Syndrome Score | the outcome will be assessed at baseline (day zero)
  The outcome measure suitable for evaluating the severity of medial tibial stress syndrome
Post-Medial Tibial Stress Syndrome Score | the outcome will be assessed after the 4 weeks.
  The outcome measure suitable for evaluating the severity of medial tibial stress syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Tahir Ramzan, Principal Investigator — Shifa Tameer-e-Millat University
Locations (1):
- Military Academy, Abbottābād, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yates B, White S. The incidence and risk factors in the development of medial tibial stress syndrome among naval recruits. Am J Sports Med. 2004 Apr-May;32(3):772-80. doi: 10.1177/0095399703258776. PMID 15090396